CLINICAL TRIAL: NCT00605150
Title: A Humanitarian Device Exemption (HDE) Use Protocol of TheraSphere for Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: HDE Use Protocol of TheraSphere for Treatment of Unresectable HCC
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: HDE# 980006
Record Dates: First submitted 2008-01-16; First posted 2008-01-30 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2022-04-22 (Actual); Status verified 2019-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Unresectable HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients enrolled: Total number of patients enrolled
  Interventions: Radiation: TheraSphere-Yttrium 90 microsphere

INTERVENTIONS:
Radiation: TheraSphere-Yttrium 90 microsphere — TheraSphere is delivered to the liver via a catheter placed into the femoral artery and guided by fluoroscopy to the hepatic artery. Once the catheter is properly positioned, the physician infuses TheraSphere, which localizes preferentially in the tumor.

SUMMARY:
MDS Nordion's TheraSphere, Yttrium-90 glass microspheres has been approved as a Humanitarian device authorized by federal(USA)law for use in radiation treatment or as a neoadjuvant to surgery or transplantation in patients with unresectable hepatocellular carcinoma(HCC)who can have placement of appropriately positioned hepatic arterial catheters. Outcomes of this treatment protocol will be monitored and reported to the Carolinas HealthCare System Institutional Review Board.

DETAILED DESCRIPTION:
The objectives of this study are to provide supervised access to treatment with TheraSphere to eligible patients with Hepatocellular Carcinoma of the liver who are not surgical resection candidates and to evaluate patient experience, toxicities and overall survival associated with TheraSphere treatment.

This is an observational treatment use protocol that will provide Institutional Review Board (IRB) oversight and documentation of the clinical experience of patients undergoing treatment for liver carcinoma using TheraSphere. Participation involves no investigational or research procedures. Patients will be followed for treatment-related adverse experiences and will be monitored in accordance with institutional practices. Approximately 60 patients will be enrolled in a treatment protocol and the number may be expanded following completion of the first cohort. The total number of patients to be treated will be determined based on clinical experience and patient outcomes. There are no control subjects in this treatment protocol.

The duration of the protocol will depend on patient experience with this treatment. An initial one year approval is sought at this time. Patient experience will be evaluated continuously and if the clinicians find that the treatment provides benefits to patients, renewal of the approval will be sought after the first 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of intrahepatic carcinoma. The histopathology confirmation criterion may be waived in patients with a radiographically identifiable liver mass, known laboratory or clinical risk factors for cancer or elevated tumor markers such as alpha feta protein (AFP) markers (clinical diagnosis).
* The cancer must be unresectable.
* Eastern Cooperative Oncology Group (ECOG) Performance Status Score 0-2
* Age greater than or equal to 18
* Able to comprehend and provide written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Any pre-treatment lab findings within 15 days of treatment demonstrating: absolute granulocyte count less than or equal to 1,500/ul, platelet count less than or equal to 45,000/ul, serum creatinine greater than or equal to 3.0 mg/dl, serum bilirubin greater than or equal to 4.0 mg/dl
* Any of the following contraindications to angiography and selective visceral catheterization: history of severe allergy or intolerance to any contrast media, narcotics, sedatives, or atropine; bleeding diathesis, not correctable by usual forms of therapy; severe peripheral vascular disease that would preclude catheterization
* Portal hypertension with portal venous shunt away from the liver
* Evidence of potential delivery of greater than 16.5 milliCurie (mCi) or 30 gray (Gy) absorbed dose of radiation to the lungs on either 1) first TheraSphere administration or 2) cumulative delivery of radiation to the lungs > 30 Gy over multiple treatments.
* Evidence of any detectable Tc-99m microaggregate albumin (MAA) flow to the stomach or duodenum, after application of established angiographic techniques to stop such flow.
* Significant extrahepatic disease representing an imminent life-threatening outcome
* Severe liver dysfunction or pulmonary insufficiency
* Active uncontrolled infection
* Significant underlying medical or psychiatric illness.
* Pregnant women may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be selected from the population of patients with unresectable cancer in the liver who are referred by surgeons and medical oncologists of CarolinasHealthCare System and by other referring physicians in the geographic area for regional therapy for liver cancer. Patients to be considered for treatment under this protocol will have been referred to one of the clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2008-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Iannitti, MD, Principal Investigator — Carolinas Medical Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total number of patients treated with TheraSphere was 11.
Pre-assignment Details: Candidates were selected by the physicians for treatment with TheraSphere, patient's signed informed consent and were treated if they met the criteria for treatment using the Humanitarian Device Exemption (HDE) protocol.
Groups:
- Treatment: TheraSphere, TheraSphere-Yttrium 90 microsphere, treatment for patients with unresectable hepatocellular carcinoma (HCC)
Period: Overall Study
Arm/Group | Treatment
Started | 11 (11 started)
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- TheraSphere Treatment: Total number of patients enrolled, TheraSphere treatment
Arm/Group | TheraSphere Treatment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (8.509)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression
Description: Progression of liver cancer
Time Frame: 6 months
Population: Number of participants enrolled
Measure: Number; unit: participants
Groups:
- TheraSphere Treatment: Total number of patients enrolled TheraSphere treatment for patients with unresectable HCC
Arm/Group | TheraSphere Treatment
Number analyzed (Participants) | 11
participants | 11

2. Secondary Outcome: Number of Participants With Unacceptable Side Effects After Treatment
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | TheraSphere Treatment
Number analyzed (Participants) | 11
Participants | 0

ADVERSE EVENTS:
Groups:
- TheraSphere Treatment for Patients With Unresectable HCC: Total number of patients enrolled, TheraSphere treatment for patients with unresectable HCC
Arm/Group | TheraSphere Treatment for Patients With Unresectable HCC
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes